CLINICAL TRIAL: NCT05727579
Title: DiEtary Sodium Intake Effects on Ertugliflozin-induced Changes in GFR, reNal Oxygenation and Systemic Hemodynamics: the DESIGN Study, a Randomized, Placebo-controlled, Cross-over Study With Ertugliflozin in People With Type 2 Diabetes
Brief Title: DiEtary Sodium Intake Effects on Ertugliflozin-induced Changes in GFR, reNal Oxygenation and Systemic Hemodynamics: the DESIGN Study
Acronym: DESIGN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, D van Raalte, Dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DC2022ERTU
Record Dates: First submitted 2023-01-24; First posted 2023-02-14 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus; Diabetic Kidney Disease; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies; Hypertension

STUDY DESIGN:
Intervention Model Description: While the treatment by ertugliflozin or placebo will be blinded, the sodium interventions are open-label.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- low-sodium diet; placebo (Other)
  Interventions: Other: Salt-Diet and/or Ertugliflozin
- low-sodium diet; ertugliflozin 15 once daily (Other)
  Interventions: Other: Salt-Diet and/or Ertugliflozin
- high-sodium diet; placebo (Other)
  Interventions: Other: Salt-Diet and/or Ertugliflozin
- High-sodium diet; ertugliflozin 15 mg once daily (Other)
  Interventions: Other: Salt-Diet and/or Ertugliflozin

INTERVENTIONS:
Other: Salt-Diet and/or Ertugliflozin — The interventions consist of an determined amount of dietary sodium intake in combination with either Ertugliflozin 15mg once daily or placebo

SUMMARY:
SGLT2 inhibitors such as ertugliflozin improve blood pressure and kidney outcomes in people living with diabetes through incompletely understood mechanisms, however, not all patients treated with SGLT2 inhibition have improved outcomes. Changes in kidney sodium handling is among the mechanisms by which SGLT2 inhibition may reduce blood pressure and drive beneficial kidney outcomes. This process is heavily dependent on daily sodium intake by patients receiving SGLT2 inhibitor treatment. In this study, the effect of daily sodium intake on SGLT2-inhibitor induced physiological effect is studied, including blood pressure regulation and kidney physiology.

ELIGIBILITY:
Inclusion Criteria:

* Adults with previously diagnosed T2DM according to American Diabetes Association (ADA) criteria
* HbA1c 6.5-10%
* Age 35-80 years of age
* Overweight or obese with BMI: >25 kg/m2
* We will make every effort to enrol participants of all races/ethnicities."
* Both sexes (females must be post-menopausal; no menses >1 year; in case of doubt, Follicle-Stimulating Hormone (FSH) will be determined with cut-off defined as >31 U/L)
* Ability to provide signed and dated, written informed consent prior to any study procedures
* Estimated GFR 60-90 ml/min/1.73m2 by CKD-EPI matching the eGFR range of most participants in VERTIS-CV
* Sodium intake at baseline < 200 mmol/day
* UACR < 30 mg/mmol
* All participants need to be on a stable dose of Diabetes medication, including Metformin, SU, insulin
* All participants need to be on a stable dose of RAS inhibition

Exclusion Criteria:

History of unstable or rapidly progressing renal disease

* Estimated GFR <60 mL/min/1.73m2 or eGFR > 90 mL/min/1.73m2 determined by CKD-EPI
* UACR > 30 mg/mmol
* Current/chronic use of the following medication: SGLT2 inhibitors, TZD, GLP-1RA, glucocorticoids, immune suppressants, antimicrobial agents, chemotherapeutics, antipsychotics, tricyclic antidepressants (TCAs) and monoamine oxidase inhibitors (MAOIs). Subjects on diuretics will only be excluded when these drugs cannot be stopped for the duration of the study.
* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs) will not be allowed, unless used as incidental medication (1-2 tablets) for non-chronic indications (i.e. sports injury, headache or back ache). However, no such drug can be taken within a timeframe of 2 weeks prior to renal testing
* History of diabetic ketoacidosis (DKA) requiring medical intervention (e.g. emergency room visit and/or hospitalization) within 1 month prior to the Screening visit.
* Current urinary tract infection and active nephritis
* Recent (<6 months) history of cardiovascular disease, including:

  * Acute coronary syndrome
  * Chronic heart failure (New York Heart Association grade II-IV)
  * Stroke or transient ischemic neurologic disorder
* Severe hepatic insufficiency and/or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
* History of or actual malignancy (except basal cell carcinoma)
* History of or actual severe mental disease
* Substance abuse (alcohol: defined as >4 units/day)
* Allergy to any of the agents used in the study
* Individuals who are investigator site personnel, directly affiliated with the study, or are immediate (spouse, parent, child, or sibling, whether biological or legally adopted) family of investigator site personnel directly affiliated with the study
* Inability to understand the study protocol or give informed consent

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the modifying effect of sodium intake on Ertugliflozin on blood pressure | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on 24-hour blood pressure in overweight/obese adults with type 2 diabetes

SECONDARY OUTCOMES:
To investigate the effect of Ertugliflozin on the hypertensive effects of high dietary sodium intake | 24 weeks
  To investigate the efficacy of ertugliflozin 15 mg daily, versus placebo, in overweight/obese adults with type 2 diabetes to reduce the hypertensive effects of a high-sodium diet (250 mmol per day) versus participant's normal diet (170 mmol/per day).

OTHER OUTCOMES:
Glomerular filtration rate (GFR) | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on GFR.
Hematocrit | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on hematocrit.
Blood pressure | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on blood pressure.
Kidney oxygenation | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on kidney oxygenation.
Effective renal plasma flow | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on effective renal plasma flow.
Renal vasculare resistance | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on renal vasculare resistance.
Body anthropometrics | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on body anthropometrics
Fasting plasma glucose | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on fasting plasma glucose
Albumin excretion rate | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on albumin excretion rate
Glucose excretion | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on 24hr urinary glucose excretion
Biomarkers | 24 weeks
  To investigate the modifying effects of WHO-recommended sodium intake (90 mmol per day) vs. high sodium intake (targeted at 250 mmol per day) on the effect of ertugliflozin 15 mg daily, versus placebo, on biomarkers

IPD SHARING:
Plan to Share IPD: Undecided